CLINICAL TRIAL: NCT02552641
Title: Food Effect on the Eradication Rate of H. Pylori With Triple Therapy With Esomeprazole
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIMESO
Record Dates: First submitted 2015-09-02; First posted 2015-09-17 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Esomeprazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Test 1 (Experimental): Esomeprazole, Amoxicillin, Clarythromycin - Administration of 20 mg esomeprazole, 1 g amoxicillin, and 500 mg clarithromycin together, in fasting conditions, twice daily
  Interventions: Other: Food effect; Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarythromycin
- Test 2 (Experimental): Esomeprazole, Amoxicillin, Clarythromycin - Administration of 20 mg esomeprazole, 1 g amoxicillin, and 500 mg clarithromycin together, after meals, twice daily
  Interventions: Other: Food effect; Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarythromycin
- Test 3 (Experimental): Esomeprazole, Amoxicillin, Clarythromycin - Administration of 20 mg esomeprazole, 1 g amoxicillin, and 500 mg clarithromycin together, twice daily in schedules variables with an interval of at least 8 hours between the doses
  Interventions: Other: Food effect; Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarythromycin

INTERVENTIONS:
Other: Food effect
Drug: Esomeprazole
Drug: Amoxicillin
Drug: Clarythromycin

SUMMARY:
The purpose of the study is assess whether the various forms of triple regimen of administration of treatment of Helicobacter pylori (before meals (fasting), after meals, and any independent mealtime) influence the rate of eradication of this bacterium.

DETAILED DESCRIPTION:
Phase IV, open, randomized, prospective study.

* Length of experience: 180 days.
* 06 visits.
* Evaluation of the efficacy of differences regimens of administration.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes;
* Age greater than or equal to 18 and less than or equal to 50 years;
* Participant diagnosed with type dyspepsia epigastric pain carriers of Helicobacter pylori infection, according to the classification of ROME III;
* Ability to understand and consent to participate in this clinical study, manifested by reading, understanding and signing of the Informed Consent (IC).

Exclusion Criteria:

* Any finding of clinical observation (clinical evaluation / physical) that is interpreted by the investigator as a medical risk to participate in the clinical trial;
* Any laboratory examination found that the investigator doctor considers a risk to the research participant for their participation in the clinical trial;
* Known hypersensitivity to the drug components used during the study;
* Women in pregnancy or breastfeeding period;
* Women in reproductive age who do not agree to use acceptable methods of contraception (oral contraceptives, injectable contraceptive, IUD, hormonal implants, barrier methods, abstinence, hormonal patch and tubal ligation); except surgically sterile (bilateral oophorectomy or hysterectomy);
* Participating in the research that has participated in clinical trial protocols in the last twelve (12) months (CNS Resolution 251 of August 7, 1997, Part III, sub-item J), unless the investigator considers that there may be direct benefit to it;
* Party that has some kinship to the second degree or bond with employees or employees of Sponsor and Research Center;
* Patients with predominant symptoms of reflux or irritable bowel syndrome, warning symptoms, peptic ulcer history or previous surgery in the upper segment of the gastrointestinal tract;
* Patients with prior treatment history of eradication of Helicobacter pylori;
* Patients with kidney, liver or heart failure;
* Patients with past or current history of alcohol abuse;
* Patients with a history of use of antibiotics or bismuth in the 4 weeks prior to study entry, PPIs or H2 blockers, NSAIDs or aspirin in the last two weeks;
* Patients whose endoscopy show changes except hyperemic gastritis, erosive gastritis den considering the maximum of 5 erosions in this location or hiatal hernia;
* Patients whose ultrasonography show hepato-biliopancreatic changes except steatosis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-02 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Rate of H pylori eradication | 7 days

SECONDARY OUTCOMES:
side effects in each of the forms of triple therapy administration and compare them | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Decio Chinzon, Phd, Principal Investigator — University of Sao Paulo
Locations (1):
- Universidade de São Paulo, São Paulo, Brazil